CLINICAL TRIAL: NCT04360798
Title: The Comparison of the Effectiveness of Unilateral and Bilateral Exercise Training in Patients With Lateral Ankle Instability
Brief Title: The Effectiveness of Unilateral and Bilateral Exercise Training in Patients With Lateral Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Burcu Pamukçu, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bpamukcu
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Chronic Ankle Instability
Keywords: Lateral Ankle Instability; Unilateral Exercise; Billateral Exercise; Ankle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral Exercise Group (Experimental): The group to which exercise protocol consisting of strengthening, stretching, range of motion, static and dynamic postural control exercises will only be applied to the affected lower extremities of the participants.
  Interventions: Other: Unilateral Exercise Group
- Bilateral Exercise Group (Experimental): The group to which exercise protocol consisting of strengthening, stretching, range of motion, static and dynamic postural control exercises will be applied to the both lower extremities of the participants.
  Interventions: Other: Bilateral Exercise Group

INTERVENTIONS:
Other: Unilateral Exercise Group — Exercise programs will be practiced 60 days, 2 days a week for 4 weeks. The entire exercise protocol will be carried out under the supervision of a physiotherapist. During the treatment session, participants exercises will only be done for 60 minutes with the affected lower extremities.
  Arms: Unilateral Exercise Group
Other: Bilateral Exercise Group — Exercise programs will be practiced 60 days, 2 days a week for 4 weeks. The entire exercise protocol will be carried out under the supervision of a physiotherapist. During the treatment session, participants will complete their exercises with both lower extremities for 30 minutes.
  Arms: Bilateral Exercise Group

SUMMARY:
70% of the general population suffers ankle injuries at least once in their lifetime. The ankle lateral ligament injuries cause an average of 6.9 days of work loss, and it has been reported that the quality of life of these patients is affected by their long-term results. Exercise training is important to prevent job loss, increase individuals' quality of life, or speed up their return to work. Functional or chronic insufficiency resulting from ankle ligament injury results in various abnormalities in the lower extremity. Motor coordination disorders due to instability, adhesions, peroneal muscle weakness, and loss of proprioception can be seen in the talus or subtalar joint. Instabilities are usually caused by loss of strength after an acute lateral ligament injury, hypomobility in the joint, inadequate improvement in proprioception, or inadequate healing of the ligament.

Almost 40% of patients with lateral ankle injury develop a condition known as chronic ankle instability. The cause of chronic ankle instability is classified as mechanical ankle instability (MAI) and functional ankle instability (FAI). While MAI is caused by ligament laxity, other factors such as proprioceptive problems, neuromuscular problems, postural control deficiencies, and muscle weakness are caused by FAI. For this reason, peroneal muscle strengthening, Achilles tendon stretching, balance training, and proprioceptive training are shown as the most important components of the treatment program in the rehabilitation of ankle instabilities. (5) It has been reported by many researchers that functional instability can be reduced and repetitive injuries can be prevented in patients given proprioceptive training and peroneal muscle strengthening on the balance board. In the results of another study evaluating bilaterally in the lower limb after balance training given to the intact side in individuals with chronic ankle instability, it was stated that the balance function of the unstable ankle was developed.

Although the treatment methods of ankle instability vary, there are very limited studies comparing treatment methods unilaterally and bilaterally in the ankle lateral instability in the literature. Our study will contribute to the literature to the next rehabilitation programs by comparing unilateral and bilateral exercise training prepared by rehabilitation protocols in many ways in two different groups.

DETAILED DESCRIPTION:
Ankle ligament injuries are one of the most common musculoskeletal injuries among physically active people, accounting for ~ 14% of all sports-related orthopedic clinic visits. And it is stated that injuries that delay the return to sports the most. 4% of these injuries and the most common are the lateral ankle ligament injuries. 70% of the general population, not only specific to sports, suffers ankle injuries at least once in their lifetime. The ankle lateral ligament injuries cause an average of 6.9 days of work loss, and it has been reported that the quality of life of these patients is affected by their long-term results. When people who play sports are taken into consideration, an ankle sprain can affect the quality of life of the individual, as well as reduce performance and keep it away from education and competition.

Ankle sprains often occur during physical activities such as basketball and football, which require sudden stops, bounces, landings, and swings around a stable foot. Most lateral ankle sprains occur when combined with excessive inversion or adduction with additional plantar flexion.

Functional or chronic deficiencies develop in the lower limbs as a result of ankle ligament injury, resulting in various abnormalities. Motor coordination disorders due to instability, adhesions, peroneal muscle weakness, and loss of proprioception can be seen in the talus or subtalar joint. Instabilities are usually caused by loss of strength after an acute lateral ligament injury, hypomobility in the joint, inadequate improvement in proprioception, or inadequate healing of the ligament. Almost 40% of patients with lateral ankle injury develop a condition known as chronic ankle instability (CAI). CAI is characterized by the occurrence of recurrent cases of instability that cause constant ankle sprain and the giving-way sensation of the ankle after the first ankle sprain. The diagnostic criteria are detailed in the International Ankle Consortium, Cumberland Ankle Instability Tool (CAIT) is often used to evaluate functional ankle instability.

Among the most important factors causing instability in the ankle are proprioceptive disorders, pain, and muscle weakness. Therefore, rehabilitation programs generally focus on exercises that include muscle strengthening, balance training, neuromuscular training, and proprioceptive training protocols. In another combined supporting study, Huang et al. investigated the effects of combined balance exercises with plyometric exercise against plyometric exercise in individuals with functional ankle instability and showed that the combined program will reduce postural oscillation in static conditions, and improve stability and energy propagation models in dynamic postural control. One of the factors contributing to CAI is thought to be the loss of strength of the ankle circumference muscle groups in both concentric and eccentric directions. It is assumed that a decrease in the strength of the muscles of the more proximal joints, such as knee and hip, not just ankle oriented, may also be effective in the formation of CAI.

It has been shown in systematic review and meta-analysis that proprioception disorder contributes to chronic ankle imbalance. In another study in individuals with unilateral chronic ankle instability, both extremities were evaluated in terms of strength and proprioception, a decrease in the sensation of kinesthesia was observed, and loss of eversion force and proprioceptive disorders were reported on both sides.

Although ankle instability treatment approaches vary widely in all these studies, there is no detailed study comparing applications unilaterally and bilaterally in the literature. Our study will contribute to the literature to the next rehabilitation programs by comparing unilateral and bilateral exercise training prepared by rehabilitation protocols in many ways in two different groups

ELIGIBILITY:
Inclusion Criteria:

* Being a volunteer between the ages of 18-45
* Mild (grade I), Moderate (grade II) or severe (grade III) lateral ankle sprain
* Ability to understand and apply Turkish written and verbal instructions.

Exclusion Criteria:

* Being an athlete
* Previous surgical interventions for the musculoskeletal system structure on both lower extremities
* History of fractures in both lower extremities
* Acute injury of musculoskeletal structures of other lower limb joints in the past 3 months
* Presence of chronic pain and edema in the foot or ankle unrelated to sprains
* Presence of other lower extremity injuries
* To have received a physiotherapy and rehabilitation program in the last 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure | 2 weeks
  The Foot and Ankle Ability Measure (FAAM) is a self-report outcome instrument developed to assess physical function for individuals with foot and ankle related impairments.The Foot and Ankle Ability Measure is a 29-item questionnaire divided into two subscales: the Foot and Ankle Ability Measure, 21-item Activities of Daily Living Subscale and the Foot and Ankle Ability Measure, 8-item Sports Subscale. The Sports subscale assesses more difficult tasks that are essential to sport, it is a population-specific subscale designed for athlete
Visual Analog Scale | 2 weeks
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.[1] It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. The pain VAS is a unidimensional measure of pain intensity, which has been widely used in diverse adult populations.
Single Heel Rise Test | 2 weeks
  It is used to test the muscle strength of the ankle plantar flexors. The participants will be asked to repeat the movement until the point they cannot perform due to pain or fatigue, and their repetition numbers will be noted. In the test, the number of 25 repeats is considered normal.
Single Leg Stance Test | 2 weeks
  Single Leg Stance Test is used to measure static balance. The person is asked to stand on one leg for 60 seconds.
  The time it remains in balance is recorded. Contact of the leg in the air with any surface is considered unsuccessful. It is applied in two different ways: eyes open and eyes closed.
Assesment of Lower Limb Muscle Strength | 2 weeks
  Hand held dynamometer, which is a valid and reliable method, will be used to evaluate the muscle strength of the lower limbs. Plantar flexion, dorsiflexion inversion and eversion muscle strength, hip flexion, extension, abduction, adduction, internal rotation and external rotation muscle strength of the participants will be measured. The highest value obtained by performing 3 attempts in each measurement will be recorded.
Balance Error Scoring System | 2 weeks
  The Balance Error Scoring System is an objective measure of assessing static postural stability. In the evaluations, 2 different surfaces are used, one of which is hard and the other is soft ground. .Postural stability is evaluated for 20 seconds in 3 different positions as double foot, single foot and tandem posture on each floor. Scoring is done according to the number of errors made. The lowest score is 0 errors and the highest score is 6. Points from the subcategory are added to calculate the total score.
Star Excursion Balance Test | 2 weeks
  It is used to evaluate the dynamic balance and postural control of the participants. The test layout consists of 8 lines arranged at a 45 ° angle from a center point. Participants will be asked to reach as much as possible in 8 different directions with one leg while standing in balance with one leg. The distance reached is recorded.
Joint Position Sensation Measurement | 2 weeks
  The perception of the joint position is measured by active and passive repositioning.
  Passive repositioning: The person to be tested is asked to learn the position by positioning the joint at a certain angle. Then, when the joint is passively moved, it is asked to stop the movement when it reaches the previously learned position. The numerical difference between the angle the person finds and the angle previously taught is evaluated.
  Active repositioning: The person who was previously taught to find the position taught by the person is asked to move and the numerical difference is recorded.
Vertical Jump Test | 2 weeks
  The Vertical Jump (Sargent Jump) test is used to assess the person's vertical explosive force. In the test, the maximum height that the person can reach by lifting his arm while standing still is measured. Then the person is asked to jump as high as he can reach where he is. In the evaluation, the difference between the height that the individual can reach when standing and the height that he can reach by jumping is taken. This test is repeated three times, the best of all jumps are the performance of the person.
Single Leg Jumping Distance Measurement | 2 weeks
  Single Leg Jump test is a valid and reliable functional performance test where participants are asked to jump forward as much as possible (53). The distance between the jump is measured by reference to the toes.
Side jump Test | 2 weeks
  Participants are asked to jump 30 cm on one leg. It consists of jumping up to 30 cm again and returning to the starting point. Each participant is asked to repeat 10 times and do it as quickly as possible. Completion time is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Univercity-Cerrahpasa, Istanbul, Turkey (Türkiye)